CLINICAL TRIAL: NCT06910410
Title: An App to Disrupt the Link Between Social Media and Negative Body Image And Disordered Eating: A Pilot Study Of Feasibility, Acceptability, and Preliminary Efficacy
Brief Title: An App to Reduce Social Media's Impact on Body Image and Eating Disorders
Acronym: BodyScreen
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Sandra Meier, Associate Professor, Dalhousie University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BODYSCREEN
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Anorexia Nervosa; Bulimia; Body Dissatisfaction; Self-esteem; Perfectionism; Disordered Eating Behaviors
Keywords: self-esteem; perfectionism; disordered eating; youth mental health
MeSH Terms: conditions — Anorexia Nervosa; Bulimia; Disordered Eating Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BodyScreen App Arm (Experimental): All participants will receive the BodyScreen app intervention. Participants will complete daily self-esteem exercises such as reflection, affirmations, challenging negative self-talk, perfectionism and low body-image.
  Interventions: Behavioral: BodyScreen App

INTERVENTIONS:
Behavioral: BodyScreen App — The BodyScreen App uses behavioural interventions along with haptic interruptions in social media app usage. The app will engage participants by sending them notifications, reminders, and activities to complete throughout the day and the week.

SUMMARY:
Social media (SM) is a key communication tool, particularly for young women aged 15-29. While SM fosters social connections, it is also linked to negative effects on mental health, including poor body image, low self-esteem, and maladaptive perfectionism. These issues arise due to social comparison with idealized images, especially on platforms like Instagram, which can contribute to disordered eating behaviours. Research suggests that reducing SM use can improve mental well-being, body image, and eating disorder symptoms. However, current interventions have not simultaneously addressed both reducing SM exposure and strengthening protective psychological factors. To address this gap, the proposed study aims to pilot BodyScreen, an intervention app designed to limit SM exposure while enhancing self-esteem and reducing perfectionism in young women at high risk for eating disorders. The study hypothesizes that BodyScreen will be feasible, acceptable, and effective in improving body image, self-esteem, and SM use, with sustained benefits at a 3-month follow-up. The intervention includes a virtual face-to-face session, mid-intervention email support, and a four-week app-based program using Ecological Momentary Interventions (EMIs). Participants will receive reminders to complete exercises designed to improve self-perception and reduce the negative effects of SM. Additionally, Ecological Momentary Assessment (EMA) will track real-time self-esteem, perfectionism, and body image, while mobile sensing will monitor SM use to tailor interactive exercises accordingly. By integrating exposure reduction with psychological strengthening, BodyScreen aims to provide a novel, evidence-based approach to mitigating the harmful effects of SM on young women's mental health.

DETAILED DESCRIPTION:
The investigators will recruit a total of 50 women, aged 15-29 years, at high risk for eating disorders to take part in a 4-week daily EMI. Participants will be recruited via advertisements placed online via social media (e.g. Instagram, Facebook, Kijiji); in print, at local universities, schools, hospitals, museums, and healthcare settings; and through participant databanks in Halifax and Toronto. This two-center design will facilitate recruitment, data collection, and generalizability, as well as preparation for a future multiple-site randomized clinical trial (RCT). These methods have previously resulted in recruiting 10-15 women per month to RCTs run by Dr. Meier's laboratory alone. Consistent with the investigator's previous research, recruitment will be tailored to promote inclusivity of sexually and racially diverse women. Yet given the differences in liability to negative body image, disordered eating and SM use, the current pilot study will focus on women only. Potential participants will be invited to complete screening questions and those who are eligible at screening will be invited to proceed to the consent process. Answers will be immediately assessed by the study website using pre-defined acceptance criteria. Participants will then receive an immediate, on-screen message stating their eligibility status to continue as a participant in the study. Ineligible participants will be informed that they do not meet the study's requirements, thanked for their interest in participating, and encouraged to take part in future PROSIT studies. Those who are eligible will be invited to continue to complete consent forms. Screening and consent will be carried out using REDCap. Participants will be emailed a link to the appropriate consent form through the "REDCap" system. During online Consent, the participant will be taken through a series of sections on the website that describes what it means to participate (e.g., reiterating the right to withdraw from the study at any time) and at the end of the consent form, participants will be asked questions (i.e. true/false and yes/no) regarding the form's contents to ensure they have correctly understood the information before proceeding that they understand the study, its risks and benefits, and/or have any questions. Participants will be encouraged to contact the research staff if they have any questions regarding the study, and all questions will be answered to their satisfaction. The script is designed to give potential study participants ample time to make an informed decision about participation. The "REDCap" recruitment site will record the date and time that online Consent, along with a space for their signature. If online Consent is submitted by participants meeting the study criteria, the "REDCap" recruitment system will automatically send an email Consent Confirmation to the participants for their records. This original document will be placed in the participant's file. Once participants have submitted confirmation of consent, the Research Assistant will generate a participant ID. After the participant ID is created, the Research Assistant will email the participants with a secure link and login with instructions on how to complete the study's online questionnaires and how to download the app. Online Consent will take <15 mins. Outcome measures will be administered using the secure online survey platform (REDCap). All scales that have been selected have robust psychometric properties, good reliability and validity. At baseline, participants will report their age, sexual orientation, socioeconomic status, educational attainment, and race/ethnicity, only at baseline using the demographic questionnaire. The proposed study's primary outcomes will be body image and eating disorder symptomology, which will be assessed with the Eating Disorder Risk Composite (EDRC) score (Eating Disorder Inventory-3; EDI-3). Secondary and tertiary outcomes for this study will be self-esteem and perfectionism, which will be assessed using the 10-item Rosenberg Self-Esteem Scale (RSES) and the 45-item Big Three Perfectionism Scale (BTPS), respectively. These assessments - EDI-3, RSES, BTPS - will be administered to participants pre- and post-intervention, as well as at the 3-month follow-up. The BodyScreen app will be used to record completed EMI exercises and allow participants to report technical issues, and SM via mobile sensing. Post-intervention, all participants will be asked to self-report the usability of the app using the System Usability Scale (SUS) adapted for digital health apps on a 5-point Likert scale. Additionally, ten participants will be invited for a semi-structured interview, conducted online or in person, depending on preference, to provide more detailed feedback and suggestions on app layout, design, and usability. While participants are using the app, the app will passively record their screen time using the phone's built-in screen and app logs. For app usage, the investigators will record the name of the app, duration, and time of usage will be recorded. During the 4 weeks of the intervention, participants will also complete EMAs three times every other day to assess momentary self-esteem, perfectionism, and body image. All data will be stored on the investigator's secure servers at Dalhousie University and the IWK Health Center using SSL connections to prevent third parties' interception. Uploads will occur daily when the device is plugged in and connected to Wi-Fi.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 15-29 years old
* Ability to provide informed consent
* Access to a smartphone (iOS or Android)
* A score greater than 47 on the Eating Disorder Risk Composite (EDRC) from the Eating Disorder Inventory-3 (EDI-3) is considered to be at high risk for an eating disorder and therefore makes a participant eligible for this study.
* Use of social media (SM) for appearance-related reasons.

Exclusion Criteria:

* A concurrent treatment for self-esteem, perfectionism, body image, or disordered eating, as it may interfere with the intervention under investigation and will make it difficult to attribute any symptom changes to either treatment.

Ages: 15 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants who show a reduced score on the Eating Disorder Risk Composite subscales from the Eating Disorder Inventory-3. | From enrollment to three months after completion of the study.
  The proposed study's primary outcomes will be body image and eating disorder symptomology, which will be assessed with the Eating Disorder Risk Composite (EDRC) subscales from the Eating Disorder Inventory-3 (EDI-3), drive for thinness scale, bulimia scale, and body dissatisfaction scale. Each of the three subscales has a raw score range of 0 to 24. The minimum EDRC score a participant can obtain is 0, which would indicate no eating disorder risk. The maximum EDRC score a participant can obtain is 72, where they score 24 on all three EDRC subscales. Those who score higher on the EDRC are at higher risk for eating disorders; higher scores are worse outcomes, and lower scores are better outcomes.

SECONDARY OUTCOMES:
Number of participants who show an increased score on the Rosenberg Self-Esteem Scale | From enrollment to three months after sudy completion.
  The 10-item Rosenberg Self-Esteem Scale (RSES) is our secondary outcome measure, assessing overall self-esteem. Each item is rated on a 4-point Likert scale (ranging from 0 to 3), resulting in total scores from 0 to 30. Higher scores indicate better outcomes, as they reflect greater self-esteem, confidence, and self-worth. Conversely, lower scores suggest worse outcomes, indicating lower self-esteem and potential self-doubt or negative self-perception.
Number of participants who show a lowered score on the Big Three Perfectionism Scale | From enrollment to three months after sudy completion.
  The 5-Item Big Three Perfectionism Scale (BTPS) is our tertiary outcome measure, perfectionism. Each item is rated on a 1 to 5 or 1 to 7 Likert scale, resulting in total scores ranging from 5 to 35. Higher scores indicate greater perfectionism and worse outcomes.

IPD SHARING:
Plan to Share IPD: No